CLINICAL TRIAL: NCT04376645
Title: A Comparative Assessment of Occlusal Bite Force Changes After Surgical Correction of the Increased Vertical Dimension in Mandibular Prognathism Subjects: A Prospective Clinical Trial
Brief Title: Occlusal Bite Force Changes After Surgical Correction of the Increased Vertical Dimension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Elham Abu Alhaija, Professor, Jordan University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44/2018
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Orthodontic Appliance
Keywords: bite force; mandibular prognathism; increased vertical dimension; surgical correction
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Intervention Model Description: Patients were allocated into one of 2 groups as follows: - Group 1: - Class III patients with increased vertical relationship Group 2: - Class III subjects with normal vertical relationship
Masking Description: Blinding was not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1: - Class III patients with increased vertical relationship These patients were scheduled for bimaxillary surgical procedures (Maxillary advancement and mandibular setback with posterior maxillary impaction) to correct the antero-posterior and vertical skeletal discrepancies.
  Interventions: Procedure: Mandibular Setback with maxillary impaction
- Group 2 (Experimental): Group 2: - Class III subjects with normal vertical relationship These patients were scheduled for mandibular setback surgical procedure (with no posterior maxillary impaction) to correct the antero-posterior skeletal discrepancy.
  Interventions: Procedure: Mandibular setback only

INTERVENTIONS:
Procedure: Mandibular Setback with maxillary impaction — Occlusal bite force will be measured after surgery to correct vertical disproportions
  Arms: Group 1
Procedure: Mandibular setback only — Occlusal bite force will be measured after surgery without changing vertical disproportions.
  Arms: Group 2

SUMMARY:
The aim of this study was to record the OBF changes after surgical correction of mandibular prognathism in patients with or without increased vertical skeletal dimensions at different time intervals (T0: before surgery; T1: at debond; T2: 3 months post-retention).

DETAILED DESCRIPTION:
Forty-two patients who presented to orthodontic clinics with severe Class III skeletal malocclusion and were already into orthodontic preparation for orthognathic surgery were selected to participate in thestudy.

Patients were allocated into one of 2 groups as follows: - Group 1: - Class III patients with increased vertical relationship Included 22 patients (8 males, 14 females).These patients were scheduled for bimaxillary surgical procedures (Maxillary advancement and mandibular setback with posterior maxillary impaction) to correct the antero-posterior and vertical skeletal discrepancies.

Group 2: - Class III subjects with normal vertical relationship Included 20 patients (8 males, 12 females).These patients were scheduled for mandibular setback surgical procedure (with no posterior maxillary impaction) to correct the antero-posterior skeletal discrepancy.

Diagnostic records (orthopantomogram, lateral cephalogram, study casts, clinical photographs) were taken for all subjects before surgery. The same records were taken post surgery just before fixed orthodontic appliance debond.

The included patients were treated by orthodontic teaching staff and postgraduate residents at orthodontic clinics/JUST using pre-adjusted edgewise fixed appliance (3M Gemini Uniteks, 0.022" MBT prescription brackets).

Bite force was measured bilaterally in the first molar region using a portable occlusal force gauge (GM10, Nagano Keiki, Tokyo, Japan), that consisted of a hydraulic pressure gauge and a biting element made of a vinyl material encased in a polyethylene tube. 3 OBF measurements were recorded on each side and incisally with a 15 second rest between each bite, the average of the three readings was used. Three OBF measurements were considered in the analysis: the maximum OBF (MOBF) achieved by the subject, the averaged OBF on molars (AOBF), and the OBF at the incisal region (IOBF).

Number of teeth in contact was measured using double-sided articulation paper strips that was smeared with a thin layer of petroleum jelly prior to its' use so as to improve the visualization of the markings of the contact points that existed in a subject's intercuspal position.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥18 years
* severe skeletal class III malocclusion
* patients willing to undergo surgery
* no systematic medical conditions

Exclusion Criteria:

* poor oral hygiene
* heavily restored or endodontically treated first molars

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Occlusal bite force | 1 year
  measured bilaterally in the first molar region using a portable occlusal force gauge
Number of teeth in contact | 1 year
  measured using double-sided articulation paper strips that was smeared with a thin layer of petroleum jelly

CONTACTS AND LOCATIONS:
Overall Officials: Elham Abu Alhaija, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Faculty of Dentistry/Jordan University of Science and Technology Dental Teaching Clinics, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No